CLINICAL TRIAL: NCT07241676
Title: Early Recurrence and Futility After Curative-intent Resection of Pancreatic Ductal Adenocarcinoma
Brief Title: Early Recurrence After Surgery for Pancreatic Cancer
Acronym: POCEMON BLUE
Status: Enrolling by invitation | Type: Observational
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, Prof. Umberto Cillo, Professor, Azienda Ospedaliera di Padova
Other Study IDs: AOP3909
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC); Recurrent Pancreatic Adenocarcinoma
Keywords: pancreatic ductal adenocarcinoma; early recurrence
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Curative-intent resection cohort: Adult patients with histologically confirmed PDAC who undergo curative-intent resection (R0 or R1), with no distant metastases, including both upfront and post-neoadjuvant cases.
  Interventions: Procedure: Curative-intent resection (R0, R1)

INTERVENTIONS:
Procedure: Curative-intent resection (R0, R1) — Standard-of-care surgical resection for pancreatic ductal adenocarcinoma, as determined by the multidisciplinary team. No study-specific interventions are mandated.

SUMMARY:
The goal of this observational study is to learn about early recurrence after curative-intent surgery for pancreatic cancer. The main questions it aims to answer are:

* How often does early recurrence (within 12 months after surgery) occur?
* When does it happen, and at which anatomical sites (liver, lung, local, peritoneum)?
* How is recurrence detected (imaging or tumor markers)?

Adults with histologically confirmed pancreatic ductal adenocarcinoma who undergo curative-intent resection without distant metastases will be enrolled. Participants will be followed according to routine clinical care at each hospital, typically with imaging and CA19-9 blood tests. No study-specific interventions are required.

DETAILED DESCRIPTION:
This international, prospective, multicenter observational study aims to characterize early recurrence (ER) after curative-intent resection of pancreatic ductal adenocarcinoma (PDAC). ER is defined as recurrence occurring within 12 months following surgery.

The study will assess the incidence, timing, anatomical sites, and detection mode (radiologic vs. biochemical) of ER, as well as post-recurrence treatment patterns and short-term outcomes. Secondary aims include comparison between neoadjuvant and upfront surgery cohorts, evaluation of biochemical-only recurrence, and identification of clinical or pathological factors predictive of ER.

Consecutive eligible patients will be enrolled from high-volume pancreatic surgery centers worldwide and followed according to institutional standards of care, typically involving routine imaging and CA19-9 surveillance. Standardized data will be prospectively collected to describe recurrence patterns and post-recurrence management. No study-specific interventions are required.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically confirmed pancreatic ductal adenocarcinoma (PDAC)
* Undergoing curative-intent resection (R0 or R1)
* No evidence of distant metastasis at the time of surgery
* Availability of preoperative CA19-9 value and pancreas-protocol CT or MRI
* Ability to provide written informed consent

Exclusion Criteria:

* Withdrawal of informed consent
* Pathological diagnosis other than PDAC (e.g., neuroendocrine tumor, acinar cell carcinoma, invasive IPMN)
* Surgery performed for palliative or diagnostic purposes only
* Intraoperative discovery of unresectable disease or distant metastases
* Gross residual disease (R2 resection)
* Incomplete clinical or radiologic follow-up precluding recurrence assessment
* Absence of adequate preoperative contrast-enhanced pancreas-protocol CT or MRI preventing accurate staging and metastatic evaluation
* Interval >9 months between two consecutive follow-up visits
* Major protocol deviations or insufficient data, as judged by the site investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with histologically confirmed pancreatic ductal adenocarcinoma undergoing curative-intent resection (R0 or R1) without evidence of distant metastases at the time of surgery. Both patients treated with neoadjuvant therapy and those undergoing upfront surgery are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence, timing, mode of detection, and anatomical site of early recurrence | Within 12 months post-surgery
  Early recurrence (ER) is defined as disease recurrence occurring within 12 months after curative-intent resection (R0 or R1) for pancreatic ductal adenocarcinoma. The incidence, time from surgery to recurrence, mode of detection (radiologic vs biochemical), and anatomical site (liver, lung, local, peritoneum, multiple) will be prospectively assessed.

SECONDARY OUTCOMES:
Comparison of ER patterns in patients treated with neoadjuvant therapy versus upfront surgery | 12 months post-surgery
  ER incidence, timing, detection mode, and anatomical sites will be compared between patients who received neoadjuvant therapy and those who underwent upfront surgery.
Incidence and clinical impact of biochemical-only recurrence | 12 months post-surgery
  Defined as sustained elevation of CA19-9 without radiologic evidence of disease. Clinical outcomes and management strategies in these patients will be analyzed.
Post-recurrence treatment strategies and short-term survival outcomes | From recurrence up to 24 months post-surgery
  Documentation of treatment intent (curative vs palliative) and treatment modality (e.g., chemotherapy, stereotactic body radiotherapy, surgery), with survival outcomes stratified by recurrence type and treatment approach.
Clinical and pathological predictors of early recurrence | Up to 12 months post-surgery
  Analysis of demographic, clinical, treatment-related, and pathological factors associated with ER to identify predictors for risk stratification and future surveillance planning.
Validation of futility criteria for upfront surgery patients | Within 6 months post-surgery
  Validation of the MetroPancreas model, with futility defined as death or recurrence within 6 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Marchegiani, MD PhD, Study Chair — University of Padova; Giampaolo Perri, MD PhD, Study Director — University of Padova
Locations (1):
- University of Padova, Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: No